CLINICAL TRIAL: NCT04388839
Title: Evolutionary Inspired Therapy for Newly Diagnosed, Metastatic, Fusion Positive Rhabdomyosarcoma
Brief Title: Evolutionary Therapy for Rhabdomyosarcoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Pediatric Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-20339
Record Dates: First submitted 2020-05-11; First posted 2020-05-14 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Rhabdomyosarcoma
Keywords: Soft Tissue Cancer; Skeletal Muscle Tissue Cancer; Sarcoma
MeSH Terms: conditions — Rhabdomyosarcoma; Sarcoma | interventions — Vincristine; Cyclophosphamide; Vinorelbine; Dactinomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Arm A - First Strike (Experimental): Participants will receive 42 weeks of conventional doses of vinorelbine, actinomycin D and cyclophosphamide
  Interventions: Drug: Cyclophosphamide; Drug: Vinorelbine; Drug: Actinomycin D
- Arm B - Second Strike - Maintenance (Experimental): Participants will receive conventional doses of Vincristine/Actinomycin D/Cyclophosphamide (VAC) until complete response (CR) for 12-42 weeks and then switch to up to 2 years of vinorelbine/oral cyclophoshamide
  Interventions: Drug: Vincristine; Drug: Cyclophosphamide; Drug: Vinorelbine; Drug: Actinomycin D; Drug: Cyclophosphamide Pill
- Arm C - Adaptive Therapy (Experimental): Therapy with VAC that starts and stops based on response, adaptive timing of therapy, with a prolonged time to progression rather than complete remission goal
  Interventions: Drug: Vincristine; Drug: Cyclophosphamide; Drug: Actinomycin D
- Arm - D Conventional Therapy (Active Comparator): Participants will receive a chemotherapy combination based on published trials. An example would be 42 weeks of VAC but may also include irinotecan, doxorubicin, ifosfamide, etoposide.
  Interventions: Drug: Vincristine; Drug: Cyclophosphamide; Drug: Actinomycin D

INTERVENTIONS:
Drug: Vincristine — IV push over 1 minute with dosing ranging from 0.24mg up to 1.5mg
  Arms: Arm - D Conventional Therapy; Arm B - Second Strike - Maintenance; Arm C - Adaptive Therapy
Drug: Cyclophosphamide — IV over 60 minutes with dosing ranging from 220mg to 1200mg
Drug: Vinorelbine — IV push over 6-10 minutes with dosing ranging from 4mg-25mg
  Other Names: Navelbine
  Arms: Arm A - First Strike; Arm B - Second Strike - Maintenance
Drug: Actinomycin D — Actinomycin D should not be given with radiation. Will be administered through IV over 3-5 minutes with dosing ranging from 0.025mg-0.045mg
  Other Names: Cosmegen
Drug: Cyclophosphamide Pill — Based on Body Surface Area (BSA) round to nearest 25mg
  Arms: Arm B - Second Strike - Maintenance

SUMMARY:
This clinical trial will evaluate 4 different strategies of chemotherapy schedules in newly diagnosed participants with metastatic Fusion Positive (alveolar) Rhabdomyosarcoma. The participant and their physician will choose from: Arm A) a first strike therapy, Arm B) a first strike-second strike (maintenance) therapy, Arm C) an adaptively timed therapy, and Arm D) conventional chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a new histologic diagnosis of rhabdomyosarcoma
* Participants must have FISH, PCR or other molecular confirmation of PAX/FOXO1 fusion per institutional standards
* Participants must have sufficient tissue (up to 10 unstained FFPE) for correlative testing
* All participants must have distant metastatic disease; either biopsy positive or PET avid extranodal or distant nodal lesions determined by the investigator to be metastatic disease. Patients with a single distant metastatic site that has been excised prior to study entry are eligible
* No prior systemic chemotherapy
* Participants enrolled to Arm B, maintenance, must be able to take oral cyclophosphamide. Note: enteral administration of cyclophosphamide is allowable.
* Males and females of reproductive potential may not participate unless they have agreed to the use of, at minimum, two methods of contraception during and after treatment or abstinence.
* Women of childbearing potential should adhere to contraception for a period of 4 months after completion of systematic chemotherapy administration
* Men who are sexually active with women of child bearing potential should adhere to contraception for a period of 4 months after completion of systematic chemotherapy administration
* All patients and/or their parents or legal guardians must have the ability to understand and the willingness to sign a written informed consent or assent document.

Exclusion Criteria:

* Participants with regional lymph nodes as the only site of disease are not eligible. Distant nodal sites alone are eligible
* Participants who are receiving any other investigational agents for rhabdomyosarcoma are ineligible
* Participants must not be receiving any additional medicines being given for the specific purpose of treating cancer. Alternative medications including, but not limited to cannabis based products would not be a reason for exclusion
* Participants are ineligible if they have uncontrolled intercurrent illness including, but not limited to:

  * ongoing or active infection not expected to resolve with current antibiotic plan
  * cardiac arrhythmia
  * psychiatric illness/social situations that would limit compliance with study requirements
* Patients who are pregnant or breastfeeding are not eligible because there is no available information regarding human fetal or teratogenic toxicities. Females of childbearing potential must have a negative serum or urine pregnancy test within 24 hours of starting protocol therapy.
* Participants who are considered unable to comply with the safety monitoring requirements of the study are not eligible

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-12-29 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
First Strike Event Free Survival | Baseline to 3 years
  Participants who choose the first strike treatment will have event free survival assessed at 3 years after initiating treatment. Event free survival is defined as time from treatment initiation to event which includes (1) any recurrence (local or regional, or distant) and (2) death due to any cause.
Second Strike Event Free Survival | Baseline to 3 years
  Participants who choose the second strike treatment will have event free survival assessed at 3 years after initiating treatment. Event free survival is defined as time from treatment initiation to event which includes (1) any recurrence (local or regional, or distant) and (2) death due to any cause
Adaptive Therapy Event Free Survival | Baseline to 3 years
  Participants who choose the adaptive therapy will have event free survival assessed at 3 years after initiating treatment. Event free survival is defined as time from treatment initiation to event which includes (1) progression that does not respond to additional VAC dosing and (2) death due to any cause

SECONDARY OUTCOMES:
Overall Survival | 5 years
  The time to event endpoint of overall survival is defined as the duration of time from diagnosis to death or last follow-up, where event would be death from any cause
Treatment-related adverse events of a certain grade or higher | Baseline to 5 years
  Number of participants with treatment-related adverse events of a certain grade or higher and hematological/biochemical toxicities based on laboratory measurements as assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Metts, MD, Principal Investigator — Moffitt Cancer Center
Locations (18):
- United States (18):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Children's Hospital of Colorado, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - University of Florida, Gainesville, Florida
  - University of Miami - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Montefiore Medical Cancer Center, The Bronx, New York
  - University of North Carolina Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center, Levine Cancer Institute, Charlotte, North Carolina
  - Duke Children's Hospital, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Vanderbilt - Ingram Cancer Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - MD Anderson, Houston, Texas
  - Primary Children's Medical Center/Utah, Salt Lake City, Utah